CLINICAL TRIAL: NCT01603979
Title: A Phase 1 Open-label, Multiple Dose, Dose Escalation Study of Monoclonal Antibody AV-203 Administered in Subjects With Metastatic or Advanced Solid Tumors
Brief Title: A Phase 1 Dose Escalation Study of AV-203, an ERBB3 Inhibitory Antibody, in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV-203-12-101
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Solid Tumors
Keywords: AV203; Solid Tumors; ERBB3; Monoclonal Antibody; HER3
MeSH Terms: interventions — AV-203

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose-escalation AV-203 Monotherapy (Experimental): dose-escalation of monotherapy AV-203 (an ERBB3 inhibitory antibody) by IV every two weeks
  Interventions: Biological: AV-203

INTERVENTIONS:
Biological: AV-203 — The antibody AV-203 is a humanized immunoglobulin G1/kappa (IgG1/κ) monoclonal antibody that targets the receptor tyrosine kinase (RTK) ERBB3 and inhibits ERBB3 activities. AV-203 will be administered as a 60 to 75-minute IV infusion once every 2 weeks until disease progression or unacceptable toxicity.

SUMMARY:
This is a Phase 1, multi-center, open-label, multiple dose, dose escalation study to evaluate the safety, tolerability, dose limiting toxicities (DLTs), maximum tolerated dose (MTD) and/or Recommended Phase 2 Dose (RP2D), pharmacokinetic (PK), pharmacodynamics, and preliminary anti-tumor activity of AV-203, an ERBB3 inhibitory antibody, administered once every 2 weeks via intravenous (IV) infusion in subjects with metastatic or advanced solid tumors. Once the RP2D is determined, patients with tumor types of interest will be evaluated in an expansion cohort at the RP2D for safety and anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Histologically and/or cytologically confirmed primary diagnosis
* Metastatic or advanced solid tumor, that has recurred or progressed following standard therapies, or for which no standard therapy exists
* Must have available tumor tissue or be willing to undergo biopsy prior to enrollment
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1
* Blood Chemistry and Hematology results within defined limits

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational agent
* Current central nervous system (CNS) or leptomeningeal metastases, or history of CNS or leptomeningeal metastases.
* Significant conduction disturbance, history of a severe arrhythmia, or history of a familial arrhythmia
* Significant cardiovascular disease
* Significant thromboembolic or vascular disorders within prior 3 months
* Any other medical condition or psychiatric condition that, in the opinion of the Investigator, might interfere with the subject's participation in the trial or interfere with the interpretation of trial results
* Known history of positive results for hepatitis C, hepatitis B, or human immunodeficiency virus.
* For female subjects, pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs, SAEs and Dose-limiting Toxicities (DLTs) | Ongoing throughout study. DLTs evaluated for first cycle of therapy. 1 cycle = 28 days

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of AV-203 | pre-dose, 5 min, 15 min, 7 hr, 24 hr, 168 hr post-dose
Time to Cmax (Tmax) of AV-203 | pre-dose, 5 min, 15 min, 7 hr, 24 hr, 168 hr post-dose
Area Under Plasma Concentration (AUC) of AV-203 | pre-dose, 5 min, 15 min, 7 hr, 24 hr, 168 hr post-dose
Terminal phase half-life (t1/2) of AV-203 | pre-dose, 5 min, 15 min, 7 hr, 24 hr, 168 hr post-dose
Clearance (Cl) of AV-203 | pre-dose, 5 min, 15 min, 7 hr, 24 hr, 168 hr post-dose
Volume of Distribution (Vd) of AV-203 | pre-dose, 5 min, 15 min, 7 hr, 24 hr, 168 hr post-dose
Objective Response Rate (ORR) | Within 28 days of first dose and every 8 weeks while on study
Disease Control Rate (DCR) | Within 28 days of first dose and every 8 weeks while on study
Duration of Response (DOR) | Within 28 days of first dose and every 8 weeks while on study
Time to Progression (TTP) | Within 28 days of first dose and every 8 weeks while on study

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - AVEO Clinical Site, Scottsdale, Arizona
  - AVEO Clinical Site, Atlanta, Georgia
  - AVEO Clinical Site, San Antonio, Texas